CLINICAL TRIAL: NCT02743871
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, THIRD-PARTY OPEN, PLACEBO-CONTROLLED, DOSE ESCALATING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS AND PHARMACODYNAMICS OF SINGLE AND/OR MULTIPLE INTRAVENOUS AND/OR SUBCUTANEOUS DOSES OF PF-06817024 IN HEALTHY SUBJECTS WHO MAY BE MILDLY ATOPIC, SUBJECTS WITH CHRONIC RHINOSINUSITIS WITH NASAL POLYPS, AND SUBJECTS WITH MODERATE-SEVERE ATOPIC DERMATITIS
Brief Title: Study Of PF-06817024 In Healthy Subjects, In Patients With Chronic Rhinosinusitis With Nasal Polyps And in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C0341001
Record Dates: First submitted 2016-04-15; First posted 2016-04-19 (Estimated); Results first posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-02

CONDITIONS: Healthy; Chronic Rhinosinusitis With Nasal Polyps; Atopic Dermatitis
Keywords: FIH, Pharmacokinetics, Pharmacodynamics, Safety, Tolerability, Atopic Dermatitis, Chronic Rhinosinusitis, Nasal Polyps
MeSH Terms: conditions — Dermatitis, Atopic; Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Cohort 1 (Experimental): 10 mg of PF-06817024 or placebo
  Interventions: Biological: PF-06817024; Other: Placebo for PF-06817024
- Cohort 2 (Experimental): 30 mg of PF-06817024 or placebo
  Interventions: Biological: PF-06817024; Other: Placebo for PF-06817024
- Cohort 3 (Experimental): 100 mg of PF-06817024 or placebo
  Interventions: Biological: PF-06817024; Other: Placebo for PF-06817024
- Cohort 4 (Experimental): 300 mg of PF-06817024 or placebo
  Interventions: Biological: PF-06817024; Other: Placebo for PF-06817024
- Cohort 5 (Experimental): 1000 mg of PF-06817024 or placebo
  Interventions: Biological: PF-06817024; Other: Placebo for PF-06817024
- Cohort 6 (Experimental): 2000 mg of PF-06817024 or placebo
  Interventions: Biological: PF-06817024; Other: Placebo for PF-06817024
- Cohort 7 (Experimental): 30 mg subcutaneous dose of PF-06817024 or placebo
  Interventions: Biological: PF-06817024; Other: Placebo for PF-06817024
- Cohort 8 (Experimental): 300 mg of PF-06817024 or placebo
  Interventions: Biological: PF-06817024; Other: Placebo for PF-06817024
- Cohort 9 (Experimental): IV dose to be determined of PF-06817024 or placebo
  Interventions: Biological: PF-06817024; Other: Placebo for PF-06817024
- Cohort 10 (Experimental): PF-06817024 or placebo
  Interventions: Biological: PF-06817024; Other: Placebo for PF-06817024
- Cohort 11 (Experimental): PF-06817024 or placebo
  Interventions: Biological: PF-06817024; Other: Placebo for PF-06817024
- Cohort 12 (Experimental): PF-06817024 or placebo
  Interventions: Biological: PF-06817024; Other: Placebo for PF-06817024
- Cohort 13 (Experimental): PF-06817024 or placebo
  Interventions: Biological: PF-06817024; Other: Placebo for PF-06817024

INTERVENTIONS:
Biological: PF-06817024 — Subjects will be given one dose of PF-06817024 intravenously
  Arms: Cohort 1; Cohort 2; Cohort 4; Cohort 5; Cohort 6; Cohort 8; Cohort 9
Other: Placebo for PF-06817024 — Subjects will be given one dose of placebo for PF-06817024 intravenously
  Arms: Cohort 1; Cohort 2; Cohort 4; Cohort 5; Cohort 6; Cohort 8; Cohort 9
Biological: PF-06817024 — Subjects will be given one dose of PF-06817024 subcutaneously
  Arms: Cohort 7
Other: Placebo for PF-06817024 — Subjects will be given one dose of placebo for PF-06817024 subcutaneously
  Arms: Cohort 7
Biological: PF-06817024 — Subjects will be given two doses of PF-06817024 intravenously
  Arms: Cohort 3
Other: Placebo for PF-06817024 — Subjects will be given two doses of PF-06817024 intravenously
  Arms: Cohort 3
Biological: PF-06817024 — Subjects will be given 2 doses intravenously
  Arms: Cohort 10; Cohort 11; Cohort 12
Other: Placebo for PF-06817024 — Subjects will be given 2 doses intravenously
  Arms: Cohort 10; Cohort 11; Cohort 12
Biological: PF-06817024 — Subjects will be given doses of PF-06817024 intravenously
  Arms: Cohort 13
Other: Placebo for PF-06817024 — Subjects will be given doses of Placebo intravenously
  Arms: Cohort 13

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, pharmacokinetics, and pharmacodynamics of PF-06817024 in healthy volunteers, in participants with chronic rhinosinusitis, with nasal polyps and in participants with moderate-to-severe Atopic Dermatitis

DETAILED DESCRIPTION:
The purpose of the study for Part 1 is to evaluate the safety and tolerability of PF-06817024 in healthy subjects.

The purpose of the study for Part 2 is to evaluate the safety and tolerability of PF-06817024 in patients with chronic rhinosinusitis with nasal polyps.

The purpose of the study for Part 3 is to evaluate the safety and tolerability of PF-06817024 in patients with moderate-to-severe Atopic Dermatitis

ELIGIBILITY:
Inclusion Criteria

* Healthy male subjects, healthy female subjects of non-childbearing potential, 18-55 years of age (Part 1)
* Male subjects, female subjects of non-childbearing potential, female subjects of childbearing potential with documented bilateral tubal ligation (tubes tied) or bilateral salpingectomy (tubes removed), 18-65 years of age, and 2 of the following symptoms: nasal congestion/obstruction, nasal discharge, face pain/pressure,or reduction/loss of smell (Part 2)
* Male or female subjects between the ages of 18 and 75 years, inclusive with moderate-to-severe Atopic Dermatitis, agree to avoid prolonged exposure to the sun and not to use tanning booths, sun lamps, or other ultraviolet light sources during the study (Part 3)

Exclusion Criteria:

* Clinically significant diseases (cardiac, psychiatric, autoimmune, renal, etc.), positive urine drug test, fever within 7 days of dosing, active infections within 28 days of dosing (Part 1 and 2 and 3)
* History of allergic reaction to topical lidocaine, nasal surgery within 6 months (Part 2)
* Exposure to live or attenuated vaccines, have skin conditions other than Atopic Dermatitis, use of JAK inhibitors and biologics (Part 3)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (20):
  - UC Davis Dermatology, Sacramento, California
  - UC Davis CTSC Clinical Research Center, Sacramento, California
  - UC Davis Health, Sacramento, California
  - New Haven Clinical Research Unit, New Haven, Connecticut
  - Dermatology Physicians of Connecticut, Shelton, Connecticut
  - ForCare Clinical Research, Tampa, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dawes Fretzin Dermatology Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Academic Dermatology, Edina, Minnesota
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Ear, Nose & Throat Specialty Care of Minnesota, P.A., Minneapolis, Minnesota
  - Prism Research, LLC, Saint Paul, Minnesota
  - Hassman Research Institute, Berlin, New Jersey
  - Carolina Phase 1 Research, LLC, Raleigh, North Carolina
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Health Concepts, Rapid City, South Dakota
  - Lee Medical Associates, PA, San Antonio, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Danto SI, Tsamandouras N, Reddy P, Gilbert SA, Mancuso JY, Page K, Beebe JS, Peeva E, Vincent MS. Exploratory pharmacodynamics and efficacy of PF-06817024 in a Phase 1 study of patients with chronic rhinosinusitis and atopic dermatitis. Allergy Asthma Clin Immunol. 2024 Aug 30;20(1):46. doi: 10.1186/s13223-024-00894-8. PMID 39215351
- [Derived] Danto SI, Tsamandouras N, Reddy P, Gilbert S, Mancuso J, Page K, Peeva E, Vincent MS, Beebe JS. Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PF-06817024 in Healthy Participants, Participants with Chronic Rhinosinusitis with Nasal Polyps, and Participants with Atopic Dermatitis: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study. J Clin Pharmacol. 2024 May;64(5):529-543. doi: 10.1002/jcph.2360. Epub 2023 Oct 30. PMID 37772436
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0341001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 97 participants were assigned and treated in this study, with 49, 20, and 28 participants in Part 1, 2, and 3, respectively.
Groups:
- Part 1 Cohort 1: PF-06817024 10 mg Intravenously (IV) Single Dose (SD): Healthy participants who might be mildly atopic received PF-06817024 10 mg IV for a SD on Study Day 1.
- Part 1 Cohort 2: PF-06817024 30 mg IV SD: Healthy participants who might be mildly atopic received PF-06817024 30 mg IV for a SD on Study Day 1.
- Part 1 Cohort 7: PF-06817024 30 mg Subcutaneously (SC) SD: Healthy participants who might be mildly atopic received PF-06817024 30 mg SC for a SD on Study Day 1.
- Part 1 Cohort 3: PF-06817024 100 mg IV SD: Healthy participants who might be mildly atopic received PF-06817024 100 mg IV for a SD on Study Day 1.
- Part 1 Cohort 3: PF-06817024 100 mg IV Multiple Doses (MD): Healthy participants who might be mildly atopic received PF-06817024 100 mg IV for MD (2 doses, on Study Days 1 and 31/46).
- Part 1 Cohort 4: PF-06817024 300 mg IV SD: Healthy participants who might be mildly atopic received PF-06817024 300 mg IV for a SD on Study Day 1.
- Part 1 Cohort 5: PF-06817024 1000 mg IV SD: Healthy participants who might be mildly atopic received PF-06817024 1000 mg IV for a SD on Study Day 1.
- Part 1: Placebo IV SD: Healthy participants who might be mildly atopic received the matching placebo of PF-06817024 IV for a SD on Study Day 1.
- Part 1 Cohort 3: Placebo IV MD: Healthy participants who might be mildly atopic received the matching placebo of PF-06817024 IV for MD (2 doses, on Study Days 1 and 46/47).
- Part 1 Cohort 7: Placebo SC SD: Healthy participants who might be mildly atopic received the matching placebo of PF-06817024 SC for a SD on Study Day 1.
- Part 2 Cohort 8: PF-06817024 300 mg IV Chronic Rhinosinusitis With Nasal Polyps (CRSwNP): Participants with chronic rhinosinusitis with nasal polyps (CRSwNP) received PF-06817024 300 mg IV for a SD on Study Day 1.
- Part 2 Cohort 8: Placebo IV CRSwNP: Participants with CRSwNP received the matching placebo of PF-06817024 IV for a SD on Study Day 1.
- Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV Atopic Dermatitis (AD): Participants with moderate to severe AD received PF-06817024 600 mg loading dose IV on Study Day 1 followed by 3 doses of PF-06817024 300 mg IV on Study Days 29, 57, and 85.
- Part 3 Cohort 13: Placebo IV AD: Participants with moderate to severe AD received the matching placebo of PF-06817024 IV on Study Days 1, 29, 57, and 85.
Period: Overall Study
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg Intravenously (IV) Single Dose (SD) | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg Subcutaneously (SC) SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV Multiple Doses (MD) | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 1: Placebo IV SD | Part 1 Cohort 3: Placebo IV MD | Part 1 Cohort 7: Placebo SC SD | Part 2 Cohort 8: PF-06817024 300 mg IV Chronic Rhinosinusitis With Nasal Polyps (CRSwNP) | Part 2 Cohort 8: Placebo IV CRSwNP | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV Atopic Dermatitis (AD) | Part 3 Cohort 13: Placebo IV AD
Started | 6 | 6 | 6 | 3 | 4 | 6 | 6 | 8 | 2 | 2 | 11 | 9 | 20 | 8
Completed | 5 | 6 | 6 | 2 | 4 | 6 | 5 | 8 | 2 | 2 | 10 | 6 | 5 | 1
Not Completed | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 15 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 12 | 6
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study medication.
Groups:
- Part 1 Cohort 1: PF-06817024 10 mg IV SD: Healthy participants who might be mildly atopic received PF-06817024 10 mg IV for a SD on Study Day 1.
- Part 1 Cohort 7: PF-06817024 30 mg SC SD: Healthy participants who might be mildly atopic received PF-06817024 30 mg SC for a SD on Study Day 1.
- Part 1 Cohort 3: PF-06817024 100 mg IV MD: Healthy participants who might be mildly atopic received PF-06817024 100 mg IV for MD (2 doses, on Study Days 1 and 31/46).
- Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP: Participants with CRSwNP received PF-06817024 300 mg IV for a SD on Study Day 1.
- Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD: Participants with moderate to severe AD received PF-06817024 600 mg loading dose IV on Study Day 1 followed by 3 doses of PF-06817024 300 mg IV on Study Days 29, 57, and 85.
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV MD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 1: Placebo IV SD | Part 1 Cohort 3: Placebo IV MD | Part 1 Cohort 7: Placebo SC SD | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP | Part 2 Cohort 8: Placebo IV CRSwNP | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD | Part 3 Cohort 13: Placebo IV AD | Total
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 6 | 6 | 8 | 2 | 2 | 11 | 9 | 20 | 8 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (4.9) | 37.0 (10.7) | 43.2 (8.7) | 27.0 (6.1) | 26.5 (6.8) | 36.3 (7.7) | 39.8 (8.7) | 33.3 (12.0) | 23.5 (0.7) | 34.5 (4.9) | 54.4 (6.2) | 42.8 (10.7) | 38.9 (13.8) | 41.0 (17.4) | 49.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 4 | 12 | 7 | 29
  Male | 6 | 6 | 4 | 3 | 4 | 6 | 6 | 7 | 2 | 2 | 8 | 5 | 8 | 1 | 68
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 3 | 3 | 1 | 1 | 1 | 1 | 3 | 0 | 1 | 11 | 7 | 8 | 3 | 44
  Black | 4 | 2 | 2 | 2 | 1 | 4 | 3 | 3 | 2 | 1 | 0 | 1 | 9 | 3 | 37
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 4
  Other | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-causality Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) in Part 1
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation where participants administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. TEAEs were events between first dose of study drug and up to discharge from study that were absent before treatment or that worsened relative to pretreatment state. An SAE was any untoward medical occurrence at any dose that: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or results in congenital anomaly/birth defect.
Time Frame: From Study Day 1 (baseline) up to Day 421 (Cohort 1 and 2), Day 601 (Cohort 3), Day 691 (Cohort 4), Day 781 (Cohort 5), and Day 511 (Cohort 7).
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 Cohort 3: PF-06817024 30 mg SC SD: Healthy participants who might be mildly atopic received PF-06817024 30 mg SC for a SD on Study Day 1.
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 3: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV MD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 1: Placebo IV SD | Part 1 Cohort 3: Placebo IV MD | Part 1 Cohort 7: Placebo SC SD
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 6 | 6 | 8 | 2 | 2
Participants
  Number of Participants With All-Causality TEAEs | 6 | 4 | 5 | 3 | 1 | 6 | 4 | 8 | 2 | 2
  Number of Participants With All-Causality SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-Related TEAEs and SAEs in Part 1
Description: An AE was any untoward medical occurrence in a clinical investigation where participants administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. TEAEs were events between first dose of study drug and up to discharge from study that were absent before treatment or that worsened relative to pretreatment state. An SAE was any untoward medical occurrence at any dose that: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or results in congenital anomaly/birth defect. The causality of TEAEs and SAEs was determined by the investigator.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV MD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 1: Placebo IV SD | Part 1 Cohort 3: Placebo IV MD | Part 1 Cohort 7: Placebo SC SD
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 6 | 6 | 8 | 2 | 2
Participants
  Number of Participants With Treatment-Related TEAEs | 2 | 2 | 2 | 2 | 1 | 3 | 1 | 1 | 0 | 1
  Number of Participants With Treatment-Related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of All-Causality TEAEs According to Severity in Part 1
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were events between first dose of study drug and up to discharge from study that were absent before treatment or that worsened relative to pretreatment state. TEAE was assessed by the investigator according to severity; Mild: did not interfere with participant's usual function; moderate: interfered to some extent with participant's usual function; severe: interfered significantly with participant's usual function.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: Events
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV MD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 1: Placebo IV SD | Part 1 Cohort 3: Placebo IV MD | Part 1 Cohort 7: Placebo SC SD
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 6 | 6 | 8 | 2 | 2
Events
  Mild | 14 | 10 | 20 | 11 | 4 | 15 | 10 | 30 | 3 | 4
  Moderate | 2 | 2 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Permanent Discontinuation Due to TEAEs in Part 1
Description: An AE was any untoward medical occurrence in a clinical investigation where participants administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. TEAEs were events between first dose of study drug and up to discharge from study that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV MD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 1: Placebo IV SD | Part 1 Cohort 3: Placebo IV MD | Part 1 Cohort 7: Placebo SC SD
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 6 | 6 | 8 | 2 | 2
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With All-Causality TEAEs and SAEs in Part 2
Description: An AE was any untoward medical occurrence in a clinical investigation where participants administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. TEAEs were events between first dose of study drug and up to discharge from study that were absent before treatment or that worsened relative to pretreatment state. An SAE was any untoward medical occurrence at any dose that: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or results in congenital anomaly/birth defect.
Time Frame: From Study Day 1 (baseline) up to Day 691.
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP | Part 2 Cohort 8: Placebo IV CRSwNP
Number analyzed (Participants) | 11 | 9
Participants
  Number of Participants With All-Causality TEAEs | 10 | 8
  Number of Participants With All-Causality SAEs | 0 | 1

6. Primary Outcome: Number of Participants With Treatment-Related TEAEs and SAEs in Part 2
Description: as for outcome 2
Time Frame: From Study Day 1 (baseline) up to Day 691.
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP | Part 2 Cohort 8: Placebo IV CRSwNP
Number analyzed (Participants) | 11 | 9
Participants
  Number of Participants With Treatment-Related TEAEs | 5 | 3
  Number of Participants With Treatment-Related SAEs | 0 | 0

7. Primary Outcome: Number of All-Causality TEAEs According to Severity in Part 2
Description: as for outcome 3
Time Frame: From Study Day 1 (baseline) up to Day 691.
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: Events
Arm/Group | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP | Part 2 Cohort 8: Placebo IV CRSwNP
Number analyzed (Participants) | 11 | 9
Events
  Mild | 44 | 24
  Moderate | 14 | 9
  Severe | 0 | 3

8. Primary Outcome: Number of Participants With Permanent Discontinuation Due to TEAEs in Part 2
Description: as for outcome 4
Time Frame: From Study Day 1 (baseline) up to Day 691.
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP | Part 2 Cohort 8: Placebo IV CRSwNP
Number analyzed (Participants) | 11 | 9
Participants | 0 | 0

9. Primary Outcome: Number of Participants With All-Causality TEAEs and SAEs in Part 3
Description: as for outcome 5
Time Frame: From Study Day 1 (baseline) up to Day 1105.
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD | Part 3 Cohort 13: Placebo IV AD
Number analyzed (Participants) | 20 | 8
Participants
  Number of Participants With All-Causality TEAEs | 12 | 5
  Number of Participants With All-Causality SAEs | 3 | 1

10. Primary Outcome: Number of Participants With Treatment-Related TEAEs and SAEs in Part 3
Description: as for outcome 2
Time Frame: From Study Day 1 (baseline) up to Day 1105.
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD | Part 3 Cohort 13: Placebo IV AD
Number analyzed (Participants) | 20 | 8
Participants
  Number of Participants With Treatment-Related TEAEs | 5 | 0
  Number of Participants With Treatment-Related SAEs | 1 | 0

11. Primary Outcome: Number of All-Causality TEAEs According to Severity in Part 3
Description: as for outcome 3
Time Frame: From Study Day 1 (baseline) up to Day 1105.
Population: All participants who received at least 1 dose of study medication.
Measure: Number; unit: TEAEs
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD | Part 3 Cohort 13: Placebo IV AD
Number analyzed (Participants) | 20 | 8
TEAEs
  Mild | 12 | 2
  Moderate | 15 | 5
  Severe | 13 | 1

12. Primary Outcome: Number of Participants With Permanent Discontinuation Due to TEAEs in Part 3
Description: An AE was any untoward medical occurrence in a clinical investigation participants administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. TEAEs were events between first dose of study drug and up to discharge from study that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From Study Day 1 (baseline) up to Day 1105.
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD | Part 3 Cohort 13: Placebo IV AD
Number analyzed (Participants) | 20 | 8
Participants | 0 | 0

13. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities in Hematology, Chemistry, and Urinalysis in Part 1
Description: Hematology parameters included hemoglobin, hematocrit, red blood cell, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet and white blood cell count, total neutrophils, eosinophils, monocytes, basophils and lymphocytes. Chemistry parameters included blood urea nitrogen, glucose (fasting), calcium, sodium, potassium, chloride, bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein. Urine parameters included pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, microscopy. Clinical significance was judged by the investigator and those met the criteria of AE are listed here. Clinically significant laboratory abnormalities reported for at least 1 participant in the whole study are presented here.
Time Frame: Part 1 single-dose cohorts: from Study Day 1 (baseline) up to Day 211. Part 1 multiple-dose cohorts: from Study Day 1 (baseline) up to Day 241.
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV MD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 1: Placebo IV SD | Part 1 Cohort 3: Placebo IV MD | Part 1 Cohort 7: Placebo SC SD
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 6 | 6 | 8 | 2 | 2
Participants
  Blood creatine phosphokinase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Transaminases increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

14. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities in Hematology, Chemistry, and Urinalysis in Part 2
Description: as for outcome 13
Time Frame: Part 2: from Study Day 1 (baseline) up to Day 211.
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP | Part 2 Cohort 8: Placebo IV CRSwNP
Number analyzed (Participants) | 11 | 9
Participants
  Blood creatine phosphokinase increased | 0 | 0
  Transaminases increased | 0 | 0

15. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities in Hematology, Chemistry, and Urinalysis in Part 3
Description: as for outcome 13
Time Frame: Part 3: from Study Day 1 (baseline) up to Day 966.
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD | Part 3 Cohort 13: Placebo IV AD
Number analyzed (Participants) | 20 | 8
Participants
  Blood creatine phosphokinase increased | 0 | 0
  Transaminases increased | 1 | 0

16. Primary Outcome: Number of Participants With Vital Sign Abnormalities in Part 1
Description: Criteria for abnormality in vital signs: supine pulse rate <40 beats per minute (bpm) or >120 bpm; supine diastolic blood pressure (DBP) <50 mmHg, maximum increase or decrease from baseline of >=20 mmHg; supine systolic blood pressure (SBP) <90 mmHg, maximum increase or decrease from baseline of >=30 mmHg. Baseline was defined as the last measurement prior to the first dosing. Vital sign abnormalities reported for at least 1 participant are presented here.
Time Frame: Study Day 1 (baseline) up to end of study (Study Day 211 for Part 1 SD cohorts, and Study Day 241 for Part 1 MD cohorts).
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV MD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 1: Placebo IV SD | Part 1 Cohort 3: Placebo IV MD | Part 1 Cohort 7: Placebo SC SD
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 6 | 6 | 8 | 2 | 2
Participants
  Maximum Increase from Baseline in Supine SBP >= 30 mmHg | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Maximum Increase from Baseline in Supine DBP >= 20 mmHg | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Maximum Decrease from Baseline in Supine SBP >= 30 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Maximum Decrease from Baseline in Supine DBP >= 20 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Supine SBP <90 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  Supine DBP <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

17. Primary Outcome: Number of Participants With Vital Sign Abnormalities in Part 2
Description: Criteria for abnormality in vital signs: supine pulse rate <40 bpm or >120 bpm; supine DBP <50 mmHg, maximum increase or decrease from baseline of >=20 mmHg; supine SBP <90 mmHg, maximum increase or decrease from baseline of >=30 mmHg. Baseline was defined as the last measurement prior to the first dosing. Vital sign abnormalities reported for at least 1 participant are presented here.
Time Frame: Study Day 1 (baseline) up to end of study (Study Day 211).
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP | Part 2 Cohort 8: Placebo IV CRSwNP
Number analyzed (Participants) | 11 | 9
Participants
  Maximum Increase from Baseline in Supine SBP >= 30 mmHg | 1 | 0
  Maximum Decrease from Baseline in Supine SBP >= 30 mmHg | 2 | 0
  Supine SBP <90 mmHg | 1 | 0

18. Primary Outcome: Number of Participants With Vital Sign Abnormalities in Part 3
Description: as for outcome 17
Time Frame: Study Day 1 (baseline) up to end of study (Study Day 337).
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD | Part 3 Cohort 13: Placebo IV AD
Number analyzed (Participants) | 20 | 8
Participants
  Maximum Increase from Baseline in Supine SBP >= 30 mmHg | 1 | 0
  Maximum Increase from Baseline in Supine DBP >= 20 mmHg | 3 | 0
  Maximum Decrease from Baseline in Supine DBP >= 20 mmHg | 2 | 0
  Supine DBP <50 mmHg | 1 | 0

19. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities in Part 1
Description: ECG abnormalities criteria included: 1) maximum QTc interval adjusted according Fridericia formula (QTcF) (msec): 450<= QTcF <480, 480<= QTcF <500, and QTcF >=500; QTcF maximum increase from baseline(msec): 30<= change <60, and change >=60; 2) maximum PR interval (msec): >=300; PR increase from baseline (msec): baseline >200 with 25% increase at maximum, baseline <=200 with 50% increase at maximum; 3) maximum QRS (msec): >=140; QRS increase from baseline (msec) >=50%. Baseline was defined as the average of the last triplicate measurement prior to the first dosing. ECG abnormalities reported for at least 1 participant are presented here.
Time Frame: as for outcome 16
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV MD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 1: Placebo IV SD | Part 1 Cohort 3: Placebo IV MD | Part 1 Cohort 7: Placebo SC SD
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 6 | 6 | 8 | 2 | 2
Participants
  450 <= maximum QTcF interval (msec) <480 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  30 <= maximum QTcF interval increase from baseline (msec) <60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0

20. Primary Outcome: Number of Participants With ECG Abnormalities in Part 2
Description: as for outcome 19
Time Frame: Study Day 1 (baseline) up to end of study (Study Day 211).
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP | Part 2 Cohort 8: Placebo IV CRSwNP
Number analyzed (Participants) | 11 | 9
Participants
  450 <= maximum QTcF interval (msec) <480 | 1 | 2
  30 <= maximum QTcF interval increase from baseline (msec) <60 | 1 | 1

21. Primary Outcome: Number of Participants With ECG Abnormalities in Part 3
Description: as for outcome 19
Time Frame: Study Day 1 (baseline) up to end of study (Study Day 337).
Population: All participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD | Part 3 Cohort 13: Placebo IV AD
Number analyzed (Participants) | 20 | 8
Participants
  450 <= maximum QTcF interval (msec) <480 | 2 | 2
  30 <= maximum QTcF interval increase from baseline (msec) <60 | 5 | 2
  Maximum QTcF interval increase from baseline (msec) >=60 | 1 | 0
  Maximum QTcF interval (msec) >=500 | 0 | 1

22. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of PF-06817024 Following Single Dose in Part 1
Description: Maximum observed serum concentration (Cmax) of PF-06817024 following single dose in Part 1; Cmax was defined as the maximum observed serum concentration.
Time Frame: Pre-dose, 1, 2, 4, 8, 12, 24, 48, 72, 96 hours post dose on Day 1, and on Follow-up Days 8, 15, 32, 46, 61, 91, 121, 151, 181, 211, and at Extended Follow-Up visits (up to a maximum of 780 days/18720 hours post dose).
Population: All enrolled participants treated who had at least 1 of the pharmacokinetic (PK) parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD
Number analyzed (Participants) | 5 | 6 | 6 | 3 | 6 | 6
ug/mL | 2.879 (19) | 12.26 (20) | 2.471 (43) | 35.56 (11) | 97.49 (7) | 313.2 (17)

23. Secondary Outcome: Cmax of PF-06817024 Following Multiple Doses in Part 1
Description: Cmax was defined as the maximum observed serum concentration.
Time Frame: Pre-dose, 1, 2, 4, 8, 12, 24, 48, 72, and 96 hr post dose on Day 1, Days 8 and 15, Day 31/46 (at pre-dose, 1, 2, 4, 8, 12, 24, 48 hr), Days 61, 91, 121, 151, 181, 211, 241, at Extended Follow-Up visits (up to a maximum of 645 days/15480 hr post dose).
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1 Cohort 3: PF-06817024 100 mg IV MD
Number analyzed (Participants) | 4
ug/mL
  Day 1 | 35.35 (15)
  Day 31: number analyzed (Participants) | 1
  Day 31 | NA (NA) — Geometric mean is not reported for N<3.
  Day 46: number analyzed (Participants) | 3
  Day 46 | 41.32 (11)

24. Secondary Outcome: Cmax of PF-06817024 in Part 2
Description: Cmax was defined as the maximum observed serum concentration.
Time Frame: Pre-dose, 1, 2, 4, 8, 12, 24, and 96 hour post dose on Day 1, and Days 8, 15, 32, 61, 91, 121, 181, 211, and at Extended Follow-Up visits (up to a maximum of 690 days/16560 hours post dose).
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP
Number analyzed (Participants) | 11
ug/mL | 107.1 (15)

25. Secondary Outcome: Cmax of PF-06817024 in Part 3
Description: Cmax was defined as the maximum observed serum concentration.
Time Frame: On Day 1 (at pre-dose, 1.5, 4, and 168 hours post dose), and Days 29, 57, and 85 (at pre-dose, 1.5 and 4 hours post dose), and on Days 113, 253, 337, and Extended Follow-Up visits (up to a maximum of 882 days/21168 hours post dose on Day 85).
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD
Number analyzed (Participants) | 20
ug/mL
  Day 1 | 197.3 (36)
  Day 29: number analyzed (Participants) | 17
  Day 29 | 165.9 (36)
  Day 57: number analyzed (Participants) | 16
  Day 57 | 190.7 (39)
  Day 85: number analyzed (Participants) | 16
  Day 85 | 199.8 (37)

26. Secondary Outcome: Dose Normalized Maximum Observed Serum Concentration (Cmax[dn]) of PF-06817024 Following Single Dose in Part 1
Description: Cmax(dn) was defined as the dose normalized maximum observed serum concentration, and calculated by Cmax/Dose. Cmax was defined as the maximum observed serum concentration.
Time Frame: as for outcome 22
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL/mg
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD
Number analyzed (Participants) | 5 | 6 | 6 | 3 | 6 | 6
ug/mL/mg | 0.2879 (19) | 0.4091 (20) | 0.08230 (43) | 0.3556 (11) | 0.3249 (7) | 0.3132 (17)

27. Secondary Outcome: Cmax(dn) of PF-06817024 Following Multiple Doses in Part 1
Description: Cmax(dn) was defined as dose normalized maximum observed serum concentration, and calculated by Cmax/Dose. Cmax was defined as the maximum observed serum concentration.
Time Frame: as for outcome 23
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL/mg
Arm/Group | Part 1 Cohort 3: PF-06817024 100 mg IV MD
Number analyzed (Participants) | 4
ug/mL/mg
  Day 1 | 0.3535 (15)
  Day 31: number analyzed (Participants) | 1
  Day 31 | NA (NA) — Geometric mean is not reported for N<3.
  Day 46: number analyzed (Participants) | 3
  Day 46 | 0.4132 (11)

28. Secondary Outcome: Cmax(dn) of PF-06817024 in Part 2
Description: as for outcome 26
Time Frame: as for outcome 24
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL/mg
Arm/Group | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP
Number analyzed (Participants) | 11
ug/mL/mg | 0.3569 (15)

29. Secondary Outcome: Cmax(dn) of PF-06817024 in Part 3
Description: as for outcome 26
Time Frame: as for outcome 25
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL/mg
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD
Number analyzed (Participants) | 20
ug/mL/mg
  Day 1 | 0.3306 (36)
  Day 29: number analyzed (Participants) | 17
  Day 29 | 0.5544 (36)
  Day 57: number analyzed (Participants) | 16
  Day 57 | 0.6361 (39)
  Day 85: number analyzed (Participants) | 16
  Day 85 | 0.6663 (37)

30. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of PF-06817024 Following Single Dose in Part 1
Description: Time to reach maximum observed serum concentration (Tmax) of PF-06817024 in Part 1; Tmax was defined as time to reach maximum observed serum concentration.
Time Frame: as for outcome 22
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD
Number analyzed (Participants) | 5 | 6 | 6 | 3 | 6 | 6
Hours | 4.00 [1.95 to 4.05] | 1.76 [1.02 to 2.33] | 338 [338 to 1080] | 1.07 [1.03 to 2.75] | 2.00 [1.53 to 8.00] | 1.775 [1.53 to 4.00]

31. Secondary Outcome: Tmax of PF-06817024 Following Multiple Doses in Part 1
Description: Tmax was defined as time to reach maximum observed serum concentration.
Time Frame: as for outcome 23
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1 Cohort 3: PF-06817024 100 mg IV MD
Number analyzed (Participants) | 4
hour
  Day 1 | 2.010 [1.03 to 8.03]
  Day 31: number analyzed (Participants) | 1
  Day 31 | NA [NA to NA] — Geometric mean is not reported for N<3.
  Day 46: number analyzed (Participants) | 3
  Day 46 | 1.550 [1.53 to 2.03]

32. Secondary Outcome: Tmax of PF-06817024 in Part 2
Description: Tmax was defined as time to reach maximum observed serum concentration.
Time Frame: as for outcome 24
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP
Number analyzed (Participants) | 11
Hours | 2.00 [1.53 to 8.00]

33. Secondary Outcome: Tmax of PF-06817024 in Part 3
Description: Tmax was defined as time to reach maximum observed serum concentration.
Time Frame: as for outcome 25
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD
Number analyzed (Participants) | 20
Hours
  Day 1 | 2.03 [1.48 to 5.12]
  Day 29: number analyzed (Participants) | 17
  Day 29 | 1.70 [1.52 to 5.17]
  Day 57: number analyzed (Participants) | 16
  Day 57 | 1.75 [1.57 to 5.15]
  Day 85: number analyzed (Participants) | 16
  Day 85 | 1.76 [1.50 to 2.83]

34. Secondary Outcome: Area Under the Curve From Time Zero to Infinity Concentration (AUCinf) of PF-06817024 Following Single Dose in Part 1 and 2
Description: Area under the curve from time zero to infinity concentration (AUCinf) of PF-06817024 following single dose in Part 1 and 2; AUCinf was defined as area under the curve from time zero to infinity concentration.
Time Frame: Pre-dose, 1, 2, 4, 8, 12, 24, and 96 hour post dose on Day 1, and Days 8, 15, 32, 61, 91, 121, 181, 211, and at Extended Follow-Up visits (up to 780 days for Part 1 and 690 days for Part 2). For Part 1 only: at post-dose 48 and 72 hour, Days 46 and 151.
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP
Number analyzed (Participants) | 5 | 6 | 6 | 3 | 6 | 5 | 11
ug*hr/mL | 4384 (28) | 14640 (28) | 8646 (38) | 44460 (22) | 116700 (23) | 427100 (10) | 146200 (19)

35. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-06817024 Following Single Dose in Part 1 and 2
Description: Area under the curve from time zero to last quantifiable concentration (AUClast) of PF-06817024 following single dose in Part 1 and 2; AUClast was defined as area under the curve from time zero to last quantifiable concentration.
Time Frame: as for outcome 34
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP
Number analyzed (Participants) | 5 | 6 | 6 | 3 | 6 | 5 | 11
ug*hr/mL | 4075 (29) | 14070 (26) | 8333 (39) | 43510 (22) | 116000 (22) | 425700 (10) | 143300 (23)

36. Secondary Outcome: Area Under the Curve Within Dosing Interval (AUCtau) of PF-06817024 Following Multiple Doses in Part 1
Description: Area under the curve within dosing interval (AUCtau) of PF-06817024 following multiple doses in Part 1; AUCtau was defined as area under the curve within dosing interval. The dosing interval was 720 hours.
Time Frame: as for outcome 23
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | Part 1 Cohort 3: PF-06817024 100 mg IV MD
Number analyzed (Participants) | 4
ug*hr/mL
  Day 1 | 10580 (11)
  Day 31: number analyzed (Participants) | 1
  Day 31 | NA (NA) — Geometric mean is not reported for N<3.
  Day 46: number analyzed (Participants) | 3
  Day 46 | 16210 (15)

37. Secondary Outcome: AUCtau of PF-06817024 in Part 3
Description: AUCtau was defined as area under the curve within dosing interval. The dosing interval was 672 hours.
Time Frame: as for outcome 25
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD
Number analyzed (Participants) | 20
ug*hr/mL
  Day 1: number analyzed (Participants) | 17
  Day 1 | 58350 (31)
  Day 29: number analyzed (Participants) | 16
  Day 29 | 77550 (38)
  Day 57: number analyzed (Participants) | 14
  Day 57 | 90340 (42)
  Day 85: number analyzed (Participants) | 15
  Day 85 | 92230 (42)

38. Secondary Outcome: Dose Normalized Area Under the Curve Within Dosing Interval (AUCtau[dn]) of PF-06817024 Following Multiple Doses in Part 1
Description: Dose normalized area under the curve within dosing interval (AUCtau[dn]) of PF-06817024 following multiple doses in Part 1; AUCtau(dn) was defined as dose normalized area under the curve within dosing interval. The dosing interval was 720 hours.
Time Frame: as for outcome 23
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL/mg
Arm/Group | Part 1 Cohort 3: PF-06817024 100 mg IV MD
Number analyzed (Participants) | 4
ug*hr/mL/mg
  Day 1 | 105.8 (11)
  Day 31: number analyzed (Participants) | 1
  Day 31 | NA (NA) — Geometric mean is not reported for N<3.
  Day 46: number analyzed (Participants) | 3
  Day 46 | 162.1 (15)

39. Secondary Outcome: AUCtau(dn) of PF-06817024 Following Multiple Doses in Part 3
Description: AUCtau(dn) was defined as dose normalized area under the curve within dosing interval. The dosing interval was 672 hours.
Time Frame: as for outcome 25
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL/mg
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD
Number analyzed (Participants) | 20
ug*hr/mL/mg
  Day 1: number analyzed (Participants) | 17
  Day 1 | 97.98 (30)
  Day 29: number analyzed (Participants) | 16
  Day 29 | 259.1 (38)
  Day 57: number analyzed (Participants) | 14
  Day 57 | 301.1 (42)
  Day 85: number analyzed (Participants) | 15
  Day 85 | 307.3 (42)

40. Secondary Outcome: Average Concentration Over Dosing Interval (Cav) of PF-06817024 Following Multiple Doses in Part 1
Description: Average concentration over dosing interval (Cav) of PF-06817024 following multiple doses in Part 1; Cav was defined as average concentration over dosing interval. The dosing interval was 720 hours.
Time Frame: as for outcome 23
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1 Cohort 3: PF-06817024 100 mg IV MD
Number analyzed (Participants) | 4
ug/mL
  Day 1 | 14.70 (12)
  Day 31: number analyzed (Participants) | 1
  Day 31 | NA (NA) — Geometric mean is not reported for N<3.
  Day 46: number analyzed (Participants) | 3
  Day 46 | 22.55 (16)

41. Secondary Outcome: Cav of PF-06817024 Following Multiple Doses in Part 3
Description: Cav was defined as average concentration over dosing interval. The dosing interval was 672 hours.
Time Frame: as for outcome 25
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD
Number analyzed (Participants) | 20
ug/mL
  Day 1: number analyzed (Participants) | 17
  Day 1 | 86.78 (30)
  Day 29: number analyzed (Participants) | 16
  Day 29 | 115.4 (38)
  Day 57: number analyzed (Participants) | 14
  Day 57 | 134.4 (42)
  Day 85: number analyzed (Participants) | 15
  Day 85 | 137.2 (42)

42. Secondary Outcome: Terminal Elimination Half Life (t1/2) of PF-06817024 Following Single Dose in Part 1
Description: t1/2 was defined as terminal elimination half life, and was calculated by Loge(2)/kel, where kel was the terminal elimination phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 22
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD
Number analyzed (Participants) | 5 | 6 | 6 | 3 | 6 | 5
Days | 91.34 (14.499) | 88.88 (15.358) | 97.17 (11.189) | 83.70 (32.608) | 83.33 (20.016) | 93.90 (5.4749)

43. Secondary Outcome: t1/2 of PF-06817024 Following Multiple Doses in Part 1
Description: T1/2 of PF-06817024 following multiple doses in Part 1; t1/2 was defined as terminal elimination half life.
Time Frame: as for outcome 23
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | Part 1 Cohort 3: PF-06817024 100 mg IV MD
Number analyzed (Participants) | 4
Day
  Day 31: number analyzed (Participants) | 1
  Day 31 | NA (NA) — Geometric mean is not reported for N<3.
  Day 46: number analyzed (Participants) | 3
  Day 46 | 98.87 (5.6083)

44. Secondary Outcome: t1/2 of PF-06817024 in Part 2
Description: as for outcome 42
Time Frame: as for outcome 24
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP
Number analyzed (Participants) | 11
Days | 85.68 (11.447)

45. Secondary Outcome: t1/2 of PF-06817024 in Part 3
Description: t1/2 was defined as terminal elimination half life, and was calculated by Loge(2)/kel, where kel was the terminal elimination phase rate constant calculated by a linear regression of the log-linear concentration-time curve. For Part 3 Cohort 13: PF-06817024 600 mg + 300 mg IV AD, t1/2 of the last dose on Day 85 was reported in the table.
Time Frame: as for outcome 25
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD
Number analyzed (Participants) | 12
Days | 75.98 (15.996)

46. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-06817024 for the Subcutaneous Cohort in Part 1
Description: Apparent volume of distribution (Vz/F) of PF-06817024 for the subcutaneous cohort in Part 1; Vz/F was defined as apparent volume of distribution.
Time Frame: as for outcome 22
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Part 1 Cohort 7: PF-06817024 30 mg SC SD
Number analyzed (Participants) | 6
L | 11.60 (37)

47. Secondary Outcome: Apparent Clearance (CL/F) of PF-06817024 for the Subcutaneous Cohort in Part 1
Description: Apparent clearance (CL/F) of PF-06817024 for the subcutaneous cohort in Part 1; CL/F was defined as apparent clearance.
Time Frame: as for outcome 22
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 1 Cohort 7: PF-06817024 30 mg SC SD
Number analyzed (Participants) | 6
L/hr | 0.003470 (38)

48. Secondary Outcome: Volume of Distribution at Steady State (Vss) of PF-06817024 Following Single Intravenous Dose in Part 1 and Part 2
Description: Volume of distribution at steady state (Vss) of PF-06817024 following a single dose in Part 1 and Part 2; Vss was defined as volume of distribution at steady state.
Time Frame: as for outcome 34
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP
Number analyzed (Participants) | 5 | 6 | 3 | 6 | 5 | 11
L | 6.949 (15) | 5.929 (22) | 6.449 (19) | 6.863 (16) | 7.260 (12) | 6.250 (17)

49. Secondary Outcome: Clearance (CL) of PF-06817024 Following Single Intravenous Dose in Part 1 and Part 2
Description: CL was defined as Clearance, calculated by Dose/AUCinf. AUCinf was defined as area under the curve from time zero to infinity concentration.
Time Frame: On Day 1 at pre-dose, post-dose 1, 2, 4, 8, 12, 24, 96 hour, Day 8, 15, 32, 61, 91, 121,181, 211, 241, 331, and 421. For Part 1 only: at post-dose 48 and 72 hour, Day 46 and 151. For Part 2 only: on Day 511, 601, and 691.
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP
Number analyzed (Participants) | 5 | 6 | 3 | 6 | 5 | 11
L/hr | 0.00228 (28) | 0.00205 (28) | 0.002249 (22) | 0.002574 (23) | 0.002341 (10) | 0.002053 (19)

50. Secondary Outcome: Trough Serum Concentration (Cmin) of PF-06817024 Post Second Dose Following Multiple Doses in Part 1
Description: Trough serum concentration (Cmin) of PF-06817024 post second dose following multiple doses in Part 1; Cmin was defined as the trough serum concentration.
Time Frame: At pre-dose on Day 31 or Day 46.
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1 Cohort 3: PF-06817024 100 mg IV MD
Number analyzed (Participants) | 4
ug/mL
  Day 31: number analyzed (Participants) | 1
  Day 31 | NA (NA) — Geometric mean is not reported for N<3.
  Day 46: number analyzed (Participants) | 3
  Day 46 | 9.851 (20)

51. Secondary Outcome: Cmin of PF-06817024 Post Last Dose Following Multiple Doses in Part 3
Description: Cmin of PF-06817024 post last dose following multiple doses in Part 3; Cmin was defined as the trough serum concentration.
Time Frame: At pre dose (0 hour) on Day 85.
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD
Number analyzed (Participants) | 15
ug/mL | 81.1 (51)

52. Secondary Outcome: Accumulation Ratio for Cmax (Rac, Cmax) of PF-06817024 Post Second Dose Following Multiple Doses in Part 1
Description: Rac, Cmax was defined as accumulation ratio for Cmax, and was calculated by (Cmax on Day 31 or Day 46) / Cmax on Day 1. Cmax was defined as the maximum observed serum concentration.
Time Frame: as for outcome 23
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1 Cohort 3: PF-06817024 100 mg IV MD
Number analyzed (Participants) | 4
Ratio
  Day 31: number analyzed (Participants) | 1
  Day 31 | NA (NA) — Geometric mean is not reported for N<3.
  Day 46: number analyzed (Participants) | 3
  Day 46 | 1.106 (3)

53. Secondary Outcome: Rac, Cmax of PF-06817024 Post Last Dose Following Multiple Doses in Part 3
Description: Rac, Cmax was defined as accumulation ratio for Cmax, and was calculated by (Cmax on Day 85) / (Cmax on Day 1). Cmax was defined as the maximum observed serum concentration.
Time Frame: as for outcome 25
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD
Number analyzed (Participants) | 16
Ratio | 2.005 (24)

54. Secondary Outcome: Accumulation Ratio for AUCtau (Rac) of PF-06817024 Post Second Dose Following Multiple Doses in Part 1
Description: Rac was defined as accumulation ratio for AUCtau. AUCtau was defined as area under the curve within dosing interval. The dosing interval was 720 hours.
Time Frame: as for outcome 23
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1 Cohort 3: PF-06817024 100 mg IV MD
Number analyzed (Participants) | 4
Ratio
  Day 31: number analyzed (Participants) | 1
  Day 31 | NA (NA) — Geometric mean is not reported for N<3.
  Day 46: number analyzed (Participants) | 3
  Day 46 | 1.499 (10)

55. Secondary Outcome: Rac of PF-06817024 Post Last Dose Following Multiple Doses in Part 3
Description: Rac was defined as accumulation ratio for AUCtau. AUCtau was defined as area under the curve within dosing interval. The dosing interval was 672 hours.
Time Frame: as for outcome 25
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD
Number analyzed (Participants) | 15
Ratio | 3.163 (20)

56. Secondary Outcome: Number of Participants With Treatment-Induced Anti-Drug Antibody (ADA) Against PF-06817024 in Part 1, 2, and 3
Description: ADA was an immunogenicity endpoint. A participant had treatment-induced ADA when baseline titer was missing or negative and the participant had >=1 post-treatment positive titer.
Time Frame: Part 1 SD cohorts: baseline up to Day 780; Part 1 MD cohort: baseline up to Day 693; Part 2: baseline up to Day 692, Part 3: baseline up to Day 964.
Population: All enrolled participants who received at least 1 dose of investigational product and had at least 1 post-treatment measurement of immunogenicity parameters of interest.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV MD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 6 | 6 | 11 | 20
Participants | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1

57. Secondary Outcome: Number of Participants With Treatment-Induced Neutralizing Antibodies (NAbs) Against PF-06817024 in Part 1, 2, and 3
Description: NAb was an immunogenicity endpoint. A participant had treatment-induced NAb when baseline titer was missing or negative and the participant had >=1 post-treatment positive titer.
Time Frame: as for outcome 56
Population: as for outcome 56
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV MD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 4 | 6 | 6 | 11 | 20
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Study Day 1 (baseline) up to Day 421 (Part 1 Cohort 1 and 2), Day 601 (Part 1 Cohort 3), Day 691 (Part 1 Cohort 4), Day 781 (Part 1 Cohort 5), and Day 511 (Part 1 Cohort 7), Day 691 (Part 2 Cohort 8), Day 1105 (Part 3 Cohort 13).
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Part 1 Cohort 1: PF-06817024 10 mg IV SD | Part 1 Cohort 2: PF-06817024 30 mg IV SD | Part 1 Cohort 7: PF-06817024 30 mg SC SD | Part 1 Cohort 3: PF-06817024 100 mg IV SD | Part 1 Cohort 3: PF-06817024 100 mg IV MD | Part 1 Cohort 4: PF-06817024 300 mg IV SD | Part 1 Cohort 5: PF-06817024 1000 mg IV SD | Part 1: Placebo IV SD | Part 1 Cohort 3: Placebo IV MD | Part 1 Cohort 7: Placebo SC SD | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP | Part 2 Cohort 8: Placebo IV CRSwNP | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD | Part 3 Cohort 13: Placebo IV AD
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/3 | 0/4 | 0/6 | 0/6 | 0/8 | 0/2 | 0/2 | 0/11 | 0/9 | 0/20 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/3 | 0/4 | 0/6 | 1/6 | 0/8 | 0/2 | 0/2 | 0/11 | 1/9 | 3/20 | 1/8
Other Adverse Events (participants affected / at risk) | 6/6 | 4/6 | 5/6 | 3/3 | 1/4 | 6/6 | 4/6 | 8/8 | 2/2 | 2/2 | 10/11 | 8/9 | 8/20 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1: PF-06817024 10 mg IV SD (N=6) | Part 1 Cohort 2: PF-06817024 30 mg IV SD (N=6) | Part 1 Cohort 7: PF-06817024 30 mg SC SD (N=6) | Part 1 Cohort 3: PF-06817024 100 mg IV SD (N=3) | Part 1 Cohort 3: PF-06817024 100 mg IV MD (N=4) | Part 1 Cohort 4: PF-06817024 300 mg IV SD (N=6) | Part 1 Cohort 5: PF-06817024 1000 mg IV SD (N=6) | Part 1: Placebo IV SD (N=8) | Part 1 Cohort 3: Placebo IV MD (N=2) | Part 1 Cohort 7: Placebo SC SD (N=2) | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP (N=11) | Part 2 Cohort 8: Placebo IV CRSwNP (N=9) | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD (N=20) | Part 3 Cohort 13: Placebo IV AD (N=8)
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema impetiginous (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adenosquamous carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1: PF-06817024 10 mg IV SD (N=6) | Part 1 Cohort 2: PF-06817024 30 mg IV SD (N=6) | Part 1 Cohort 7: PF-06817024 30 mg SC SD (N=6) | Part 1 Cohort 3: PF-06817024 100 mg IV SD (N=3) | Part 1 Cohort 3: PF-06817024 100 mg IV MD (N=4) | Part 1 Cohort 4: PF-06817024 300 mg IV SD (N=6) | Part 1 Cohort 5: PF-06817024 1000 mg IV SD (N=6) | Part 1: Placebo IV SD (N=8) | Part 1 Cohort 3: Placebo IV MD (N=2) | Part 1 Cohort 7: Placebo SC SD (N=2) | Part 2 Cohort 8: PF-06817024 300 mg IV CRSwNP (N=11) | Part 2 Cohort 8: Placebo IV CRSwNP (N=9) | Part 3 Cohort 13: PF-06817024 600 mg => 300 mg IV AD (N=20) | Part 3 Cohort 13: Placebo IV AD (N=8)
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 4 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 0 | 1 | 3 | 2 | 3 | 0 | 0 | 3 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 3 | 1 | 0 | 3 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Mouth swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Therapeutic response increased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural constipation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyposmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder due to general medical condition, insomnia type (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site reaction (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dental restoration failure (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Libido increased (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Conditional aggravated (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/71/NCT02743871/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT02743871/SAP_001.pdf